CLINICAL TRIAL: NCT03711162
Title: A Phase 3, Randomized, Double-blind, Parallel-group, Placebo-controlled Multicenter Study to Evaluate the Efficacy and Safety of Two Doses of GLPG1690 in Addition to Local Standard of Care for Minimum 52 Weeks in Subjects With Idiopathic Pulmonary Fibrosis
Brief Title: A Clinical Study to Test How Effective and Safe GLPG1690 is for Subjects With Idiopathic Pulmonary Fibrosis (IPF) When Used Together With Standard of Care
Acronym: ISABELA1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The benefit-risk profile no longer supports continuing the study
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG1690-CL-303; 2018-001405-87 (EudraCT Number)
Record Dates: First submitted 2018-10-15; First posted 2018-10-18 (Actual); Results first posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — GLPG1690

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GLPG1690 600 mg (Experimental): Participants received GLPG1690 (ziritaxestat) 600 mg, film-coated tablets orally once daily (mean GLPG1690 exposure was up to 325.3 days) in addition to local standard of care. Standard of care included either pirfenidone or nintedanib at a stable dose for at least 2 months before screening, and during screening; or neither pirfenidone or nintedanib (for any reason).
  Interventions: Drug: GLPG1690
- GLPG1690 200 mg (Experimental): Participants received GLPG1690 (ziritaxestat) 200 mg as film-coated tablet for oral use once daily (mean GLPG1690 exposure was up to 356.0 days) in addition to local standard of care. Standard of care included either pirfenidone or nintedanib at a stable dose for at least 2 months before screening, and during screening; or neither pirfenidone or nintedanib (for any reason).
  Interventions: Drug: GLPG1690
- Placebo (Placebo Comparator): Participants received GLPG1690 (ziritaxestat) matching placebo tablets for oral use once daily (mean GLPG1690 exposure was up to 353.4 days) in addition to local standard of care. Standard of care included either pirfenidone or nintedanib at a stable dose for at least 2 months before screening, and during screening; or neither pirfenidone or nintedanib (for any reason).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG1690 — GLPG1690, film-coated tablets for oral use.
  Other Names: ziritaxestat
  Arms: GLPG1690 200 mg; GLPG1690 600 mg
Drug: Placebo — Matching placebo, film-coated tablets for oral use.
  Arms: Placebo

SUMMARY:
The main purpose of this study was to see how GLPG1690 works together with your current standard treatment on your lung function and IPF disease in general. The study also investigated how well GLPG1690 is tolerated (for example if you got any side effects while on study drug).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged ≥40 years on the day of signing the Informed Consent Form (ICF).
* A diagnosis of IPF within 5 years prior to the screening visit, as per applicable American Thoracic Society (ATS)/European Respiratory Society (ERS)/Japanese Respiratory Society (JRS)/Latin American Thoracic Association (ALAT) guidelines at the time of diagnosis.
* Chest high-resolution computed tomography (HRCT) historically performed within 12 months prior to the screening visit and according to the minimum requirements for IPF diagnosis by central review based on subject's HRCT only (if no lung biopsy (LB) available), or based on both HRCT and LB (with application of the different criteria in either situation). If an evaluable HRCT <12 months prior to screening is not available, an HRCT can be performed at screening to determine eligibility, according to the same requirements as the historical HRCT.
* Subjects receiving local standard of care for the treatment of IPF, defined as either pirfenidone or nintedanib at a stable dose for at least two months before screening, and during screening; or neither pirfenidone or nintedanib (for any reason). A stable dose is defined as the highest dose tolerated by the subject during those two months.
* The extent of fibrotic changes is greater than the extent of emphysema on the most recent HRCT scan (investigator-determined).
* Meeting all of the following criteria during the screening period: FVC ≥45% predicted of normal, Forced expiratory volume in 1 second (FEV1)/FVC ≥0.7, diffusing capacity of the lung for carbon monoxide (DLCO) corrected for Hb ≥30% predicted of normal.
* Estimated minimum life expectancy of at least 30 months for non IPF related disease in the opinion of the investigator.
* Male subjects and female subjects of childbearing potential agree to use highly effective contraception/preventive exposure measures from the time of first dose of investigational medicinal product (IMP) (for the male subject) or the signing of the ICF (for the female subject), during the study, and until 90 days (male) or 30 days (female) after the last dose of IMP.
* Able to walk at least 150 meters during the 6-Minute Walk Test (6MWT) at screening Visit 1; without having a contraindication to perform the 6MWT or without a condition putting the subject at risk of falling during the test (investigator's discretion). The use of a cane is allowed, the use of a stroller is not allowed at all for any condition. At Visit 2, for the oxygen titration test, resting oxygen saturation (SpO2) should be ≥88% with maximum 6 L O2/minute; during the walk, SpO2 should be ≥83% with 6 L O2/minute or ≥88% with 0, 2 or 4 L O2/minute.

Exclusion Criteria:

* History of malignancy within the past 5 years (except for carcinoma in situ of the uterine cervix, basal cell carcinoma of the skin that has been treated with no evidence of recurrence, prostate cancer that has been medically managed through active surveillance or watchful waiting, squamous cell carcinoma of the skin if fully resected, and Ductal Carcinoma In Situ).
* Clinically significant abnormalities detected on ECG of either rhythm or conduction, a QT interval corrected for heart rate using Fridericia's formula (QTcF) >450 ms, or a known long QT syndrome. Patients with implantable cardiovascular devices (e.g. pacemaker) affecting the QT interval time may be enrolled in the study based upon investigator judgment following cardiologist consultation if deemed necessary, and only after discussion with the medical monitor.
* Acute IPF exacerbation within 6 months prior to screening and/or during the screening period. The definition of an acute IPF exacerbation is as follows: Previous or concurrent diagnosis of IPF; Acute worsening or development of dyspnea typically < 1 month duration; Computed tomography with new bilateral ground-glass opacity and/or consolidation superimposed on a background pattern consistent with usual interstitial pneumonia pattern and deterioration not fully explained by cardiac failure or fluid overload.
* Lower respiratory tract infection requiring treatment within 4 weeks prior to screening and/or during the screening period.
* Interstitial lung disease associated with known primary diseases (e.g. sarcoidosis and amyloidosis), exposures (e.g. radiation, silica, asbestos, and coal dust), or drugs (e.g. amiodarone).
* Diagnosis of severe pulmonary hypertension (investigator- determined).
* Unstable cardiovascular, pulmonary (other than IPF), or other disease within 6 months prior to screening or during the screening period (e.g. acute coronary disease, heart failure, and stroke).
* Had gastric perforation within 3 months prior to screening or during screening, and/or underwent major surgery within 3 months prior to screening, during screening or have major surgery planned during the study period.
* History of nintedanib-related increase in ALT and/or AST of >5 x upper limit of the normal range (ULN) and increased susceptibility to elevated LFT; moderate to severe hepatic impairment (Child-Pugh B or C) and/or abnormal liver function test (LFT) at screening, defined as aspartate aminotransferase (AST), and/or alanine aminotransferase (ALT), and/or total bilirubin ≥1.5 x upper limit of the normal range (ULN), and/or gamma glutamyl transferase (GGT) ≥3 x ULN. Retesting is allowed once for abnormal LFT.
* Abnormal renal function defined as estimated creatinine clearance, calculated according to Cockcroft-Gault calculation (CCr) <30 mL/min. Retesting is allowed once.
* Use of any of the following therapies within 4 weeks prior to screening and during the screening period, or planned during the study: warfarin, imatinib, ambrisentan, azathioprine, cyclophosphamide, cyclosporine A, bosentan, methotrexate, sildenafil (except for occasional use), prednisone at steady dose >10 mg/day or equivalent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Study Director, MD, Study Director — Galapagos NV
Locations (132):
- United States (47):
  - Pulmonary Associates, Phoenix, Arizona
  - Mayo Clinic Arizona - PPDS, Scottsdale, Arizona
  - Atria Clinical Research - BTC - PPDS, Little Rock, Arkansas
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Respire Research, Palm Springs, California
  - University of California San Diego, San Diego, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Western Connecticut Medical Group, Danbury, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - PAB Clinical Research - ClinEdge - PPDS, Brandon, Florida
  - St. Francis Medical Institute - BTC - PPDS, Clearwater, Florida
  - North Florida/South Georgia Veterans Health System-NAVREF-PPDS, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - Advanced Pulmonary Research Institute, Loxahatchee Groves, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Pulmonary and Infections Disease Associates, Council Bluffs, Iowa
  - University of Louisville, Louisville, Kentucky
  - Tulane Medical Center, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Division of Pulmonary and Critical Care Medicine, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Dearborn, Michigan
  - Minnesota Lung Center, Minneapolis, Minnesota
  - Mayo Clinic - PPDS, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Creighton University, Omaha, Nebraska
  - University of Rochester Medical Center - PPDS, Rochester, New York
  - PulmonIx LLC, Greensboro, North Carolina
  - UC Health Department of Internal Medicine, Pulmonary, Critical Care & Sleep Medicine, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Oregon Clinic, Portland, Oregon
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Metroplex Pulmonary and Sleep Medicine Center, McKinney, Texas
  - University of Texas Health Science Center San Antonio, San Antonio, Texas
  - University of Utah Medical Care, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Western Washington Medical Group, Everett, Washington
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Australia (10):
  - Royal Adelaide Hospital, Adelaide
  - Flinders Medical Centre, Bedford Park
  - Box Hill Hospital, Box Hill
  - Corte Royal Prince Alfred Hospital, Camperdown
  - Lung Research Queensland, Chermside
  - Concord Repatriation General Hospital, Concord
  - St Vincent's Hospital Sydney, Darlinghurst
  - Austin Health, Heidelberg
  - Respiratory Clinical Trials Pty Ltd, Kent Town
  - The Alfred Hospital, Melbourne
- Belgium (5):
  - ZNA Middelheim, Antwerp
  - Hôpital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven, Leuven
  - CHU UCL Namur asbl - Site Godinne, Yvoir
- Brazil (2):
  - Irmandade Da Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Faculdade de Medicina Do ABC, Santo André
- Chile (9):
  - Hospital Clínico Regional de Concepción Dr Guillermo Grant Benavente, Concepción
  - Centro de Investigación Curico, Curicó
  - Centro Respiratorio Integral LTDA. (CENRESIN), Quillota
  - Instituto Nacional Torax, Santiago
  - Centro de Investigaciones Medicas Respiratorias CIMER, Santiago
  - Hospital Dr Sotero Del Rio, Santiago
  - Centro de Investigacion del Maule, Talca
  - Hospital Carlos Van Buren, Valparaíso
  - CINVEC- Estudos Clínicos Quinta Región Limitada, Viña del Mar
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Ostrava, Ostrava
  - Thomayerova nemocnice, Prague
  - Nemocnice Na Bulovce, Prague
- Denmark (3):
  - Aarhus Universitetshospital, Aarhus
  - Gentofte Hospital, Hellerup
  - Odense Universitetshospital, Odense
- Germany (7):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Evangelische Lungenklinik, Berlin
  - Fachkrankenhaus Coswig, Coswig
  - Medizinische Hochschule Hannover, Hanover
  - Thorax Klinik, Heidelberg
  - Universitatsklinikum Leipzig, Leipzig
  - Klinikum Rosenheim, Rosenheim
- Greece (5):
  - Sotiria Chest Hospital of Athens, Athens
  - Attikon University General Hospital, Athens
  - University General Hospital of Heraklion, Heraklion
  - University General Hospital of Larissa, Larissa
  - Georgios Papanikolaou General Hospital of Thessaloniki, Thessaloniki
- Japan (7):
  - Tenryu Hospital, Hamamatsu
  - Saiseikai Kumamoto Hospital, Kumamoto
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakai
  - Tosei General Hospital, Seto
  - Center Hospital of the National Center for Global Health and Medicine, Tokyo
  - National Hospital Organization Kyushu Medical Center, Tokyo
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama
- Peru (6):
  - Hospital Chancay y Servicios Basicos de Salud, Chancay
  - Hospital Nacional Guillermo Almenara Irigoyen ESSALUD, Lima
  - Clinica Internacional - PPDS, Lima Cercado
  - Clinica Ricardo Palma - PPDS, San Isidro
  - Clinica Providencia (Inverconsult Sociedad Anonima), San Miguel
  - Clinica San Pablo, Santiago de Surco
- Spain (8):
  - CHUVI - H.U. Alvaro Cunquerio, Vigo, Pontevedra
  - Hospital Clinical de Barcelona, Barcelona
  - Hospital Universitario de Bellvitge, Hospitalet De Llobregat, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Clinica Universidad Navarra, Pamplona
  - Hospital Universitario Marques de Valdecilla, Santander
  - Consorcio Hospital General Universitario de Valencia, Valencia
- Taiwan (4):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (4):
  - Süreyyapaşa Göğüs Hastalıkları Ve Göğüs Cerrahisi Eğitim Ve Araştırma Hastanesi, Istanbul
  - Ege Universitesi Tıp Fakultesi Hastanesi Gögus Hastalıkları Anabilim Dalı, Izmir
  - Uludag Universitesi Tıp Fakultesi Hastanesi Gögüs Hastalıkları Anabilim Dalı, Izmir
  - Mersin Üniversitesi Tıp Fakültesi Hastanesi Göğüs Hastalıkları Polikinliği, Mersin
- United Kingdom (11):
  - Birmingham Heartlands Hospital, Birmingham
  - Southmead Hospital, Bristol
  - Papworth Hospital, Cambridge
  - Castle Hill Hospital, Cottingham
  - Royal Devon and Exeter Hospital NHS Trust, Exeter
  - Aintree University Hospital NHS Foundation Trust, Liverpool
  - Royal Brompton Hospital, London
  - Wythenshawe Hospital - PPDS, Manchester
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Nottingham City Hospital, Nottingham
  - Northern General Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ford P, Kreuter M, Brown KK, Wuyts WA, Wijsenbeek M, Israel-Biet D, Hubbard R, Nathan SD, Nunes H, Penninckx B, Prasad N, Seghers I, Spagnolo P, Verbruggen N, Hirani N, Behr J, Kaner RJ, Maher TM. An adjudication algorithm for respiratory-related hospitalisation in idiopathic pulmonary fibrosis. ERJ Open Res. 2024 Jan 29;10(1):00636-2023. doi: 10.1183/23120541.00636-2023. eCollection 2024 Jan. PMID 38288082
- [Derived] Maher TM, Ford P, Brown KK, Costabel U, Cottin V, Danoff SK, Groenveld I, Helmer E, Jenkins RG, Milner J, Molenberghs G, Penninckx B, Randall MJ, Van Den Blink B, Fieuw A, Vandenrijn C, Rocak S, Seghers I, Shao L, Taneja A, Jentsch G, Watkins TR, Wuyts WA, Kreuter M, Verbruggen N, Prasad N, Wijsenbeek MS; ISABELA 1 and 2 Investigators. Ziritaxestat, a Novel Autotaxin Inhibitor, and Lung Function in Idiopathic Pulmonary Fibrosis: The ISABELA 1 and 2 Randomized Clinical Trials. JAMA. 2023 May 9;329(18):1567-1578. doi: 10.1001/jama.2023.5355. PMID 37159034
- [Derived] Maher TM, Kreuter M, Lederer DJ, Brown KK, Wuyts W, Verbruggen N, Stutvoet S, Fieuw A, Ford P, Abi-Saab W, Wijsenbeek M. Rationale, design and objectives of two phase III, randomised, placebo-controlled studies of GLPG1690, a novel autotaxin inhibitor, in idiopathic pulmonary fibrosis (ISABELA 1 and 2). BMJ Open Respir Res. 2019 May 21;6(1):e000422. doi: 10.1136/bmjresp-2019-000422. eCollection 2019. PMID 31179008

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with centrally confirmed diagnosis of idiopathic pulmonary fibrosis (IPF) were enrolled at 106 sites.
Pre-assignment Details: A total of 1116 participants were screened for the study, and 525 were randomized and 523 were treated.
Groups:
- GLPG1690 600 mg: Participants received GLPG1690 (ziritaxestat) 600 milligrams (mg), film-coated tablets orally once daily (mean GLPG1690 exposure was up to 325.3 days) in addition to local standard of care. Standard of care included either pirfenidone or nintedanib at a stable dose for at least 2 months before screening, and during screening; or neither pirfenidone or nintedanib (for any reason).
Period: Overall Study
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Started | 175 | 175 | 175
Treated | 174 | 175 | 174
Completed | 0 | 0 | 0
Not Completed | 175 | 175 | 175
Not completed — Adverse Event | 5 | 2 | 4
Not completed — Death | 11 | 7 | 8
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Study Terminated by Sponsor | 139 | 152 | 146
Not completed — Withdrawal by Subject | 17 | 10 | 10
Not completed — Miscellaneous | 1 | 2 | 2
Not completed — Not Treated | 1 | 0 | 1
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Protocol Specified Withdrawal Criteria Met | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) consisted of all randomized participants who received at least 1 dose of investigational product (IP).
Groups:
- Total: Total of all reporting groups
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo | Total
Number analyzed (Participants) | 174 | 175 | 174 | 523
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (7.2) | 70.0 (6.7) | 70.6 (7.7) | 70.0 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 28 | 92
  Male | 142 | 143 | 146 | 431
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 27 | 26 | 97
  Not Hispanic or Latino | 129 | 145 | 148 | 422
  Unknown or Not Reported | 1 | 3 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 6 | 6 | 22
  Asian | 11 | 9 | 9 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 152 | 160 | 159 | 471
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Forced Vital Capacity (FVC) [Mean (Standard Deviation); unit: mL] — FVC (in milliliter [mL]) is the maximum amount of air exhaled from lungs by a participant after taking their deepest possible breath, as measured by spirometry.
  mL | 2947.0 (820.8) | 2873.2 (815.8) | 2943.3 (738.7) | 2921.1 (791.9)

OUTCOME MEASURES:

1. Primary Outcome: Annual Rate of Decline in FVC up to Week 52
Description: FVC (in mL) is the maximum amount of air exhaled from lungs by a participant after taking their deepest possible breath, as measured by spirometry.
Time Frame: Baseline up to week 52
Population: Full Analysis Set - Efficacy (FAS-EF) included all randomized participants who received at least 1 dose of investigational product and excluded participants from the site found to have serious good clinical practice (GCP)-noncompliance issues.
Measure: Least Squares Mean (Standard Error); unit: mL/year
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 169 | 171 | 164
mL/year | -124.6 (27.15) | -173.9 (26.31) | -147.3 (26.72)
Statistical Analysis 1: Comparison: GLPG1690 600 mg vs Placebo; Test type: Superiority; p = 0.5525, Coefficient Regression Model — P-value: based on random coefficient regression model (linear slope model) on FVC values; Treatment effect determined by using estimated slopes for each treatment group on basis of time-by-treatment interaction term from the mixed model; Least square (LS) mean difference = 22.7, 95% CI 2-sided [-52.3 to 97.6], Standard Error of Mean 38.12
Statistical Analysis 2: Comparison: GLPG1690 200 mg vs Placebo; Test type: Superiority; p = 0.4776, Coefficient Regression Model — P-value: based on random coefficient regression model (linear slope model) on FVC values; Treatment effect was determined by using estimated slopes for each treatment group on basis of time-by-treatment interaction term from mixed model; LS mean difference = -26.7, 95% CI 2-sided [-100.5 to 47.1], Standard Error of Mean 37.53

2. Secondary Outcome: Percentage of Participants With Disease Progression up to Week 52
Description: Disease progression was defined as the composite occurrence of more than or equal to (>=)10 percent (%) absolute decline in percent predicted forced vital capacity (%FVC) or all-cause mortality. FVC (in mL) is the maximum amount of air exhaled from lungs by a participant after taking their deepest possible breath, as measured by spirometry.
Time Frame: Up to week 52
Population: Full Analysis Set- Efficacy
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 169 | 171 | 164
Percentage of participants | 17.8 | 18.7 | 18.3
Statistical Analysis 1: Comparison: GLPG1690 600 mg vs Placebo; Test type: Superiority; p = 0.9648, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.56 to 1.74]
Statistical Analysis 2: Comparison: GLPG1690 200 mg vs Placebo; Test type: Superiority; p = 0.8530, Regression, Logistic; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.60 to 1.84]

3. Secondary Outcome: Percentage of Participants With Respiratory-Related Hospitalization Until End of Study (EoS)
Description: Percentage of participants with respiratory related hospitalization were reported in this measure.
Time Frame: Up to EoS (week 121)
Population: Full Analysis Set- Efficacy
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 169 | 171 | 164
Percentage of participants | 9.5 | 9.4 | 9.8
Statistical Analysis 1: Comparison: GLPG1690 600 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.50 to 2.05] — Hazard ratio and 95% confidence interval originated from a Cox proportional hazards for time to respiratory-related hospitalization
Statistical Analysis 2: Comparison: GLPG1690 200 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.47 to 1.88] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change From Baseline in St.George's Respiratory Questionnaire (SGRQ) Total Score at Week 52
Description: SGRQ is a 50-item paper questionnaire designed to measure and quantify the impact of chronic respiratory disease on health-related quality of life (QOL) and well-being, split into 3 domains: symptoms score assessing the frequency and severity of respiratory symptoms (Items 1-8), activity score assessing the effects of breathlessness on mobility and physical activity (Items 11-17 and 36 to 44), and impacts score assessing the psychosocial impact of the disease (Items 9-10, 18-35 and 45-50). Each item has a specific weight.
  Domain scores = 100 * summed weights from positive items in that component/sum of maximum weights for all non-missing items in that component
  Total score = 100 * summed weights from positive items in the questionnaire/sum of maximum weights for all non-missing items in the questionnaire
  Scores were weighted such that each domain score ranged from 0 to 100 and the total score ranged from 0 to 100, with higher scores indicating the poorer health-related QOL.
Time Frame: Baseline, week 52
Population: Full Analysis Set- Efficacy
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 169 | 171 | 164
Score on a scale | 3.3 (1.41) | 4.1 (1.32) | 3.8 (1.36)
Statistical Analysis 1: Comparison: GLPG1690 600 mg vs Placebo; Test type: Superiority; p = 0.7850, Mixed Models Analysis; LS mean difference = -0.5, 95% CI 2-sided [-4.4 to 3.3] — LS mean difference (95% CI) per treatment group with treatment, time (categorical), treatment-by-time interaction, stratum and baseline SGRQ total score as fixed effects and participant as random effect
Statistical Analysis 2: Comparison: GLPG1690 200 mg vs Placebo; Test type: Superiority; p = 0.8617, Mixed Models Analysis; LS mean difference = 0.3, 95% CI 2-sided [-3.4 to 4.1] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Annual Rate of Decline in FVC Until EoS
Description: as for outcome 1
Time Frame: Baseline up to EoS (week 121)
Population: Full Analysis Set - Efficacy
Measure: Least Squares Mean (Standard Error); unit: mL/year
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 169 | 171 | 164
mL/year | -127.0 (24.01) | -175.5 (22.97) | -146.4 (23.59)
Statistical Analysis 1: Comparison: GLPG1690 600 mg vs Placebo; Test type: Superiority; LS Mean difference = 19.4, 95% CI 2-sided [-46.9 to 85.7], Standard Error of Mean 33.68 — The treatment effect was determined by using estimated slopes for each study group on the basis of the time-by-treatment interaction term from the mixed model
Statistical Analysis 2: Comparison: GLPG1690 200 mg vs Placebo; Test type: Superiority; LS Mean difference = -29.1, 95% CI 2-sided [-93.9 to 35.8], Standard Error of Mean 32.95 — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Percentage of Participants With Disease Progression Until EoS
Description: Disease progression was defined as the composite occurrence of >=10% absolute decline in percent predicted %FVC or all-cause mortality. FVC (in mL) is the maximum amount of air exhaled from lungs by a participant after taking their deepest possible breath, as measured by spirometry.
Time Frame: Up to EoS (week 121)
Population: Full Analysis Set - Efficacy
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 169 | 171 | 164
Percentage of participants | 23.1 | 24.6 | 21.3
Statistical Analysis 1: Comparison: GLPG1690 600 mg vs Placebo; Test type: Superiority; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.68 to 1.95] — Odds ratio and 95% confidence interval originated from a logistic regression
Statistical Analysis 2: Comparison: GLPG1690 200 mg vs Placebo; Test type: Superiority; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.74 to 2.09] — Odds ratio and 95% confidence interval originated from a logistic regression

7. Secondary Outcome: Change From Baseline in St.George's Respiratory Questionnaire (SGRQ) Total Score at Week 100
Description: as for outcome 4
Time Frame: Baseline, week 100
Population: Full Analysis Set - Efficacy
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 169 | 171 | 164
Score on a scale | 11.4 [0.3 to 22.6] | 10.5 [1.1 to 20.0] | 7.7 [-2.7 to 18.0]
Statistical Analysis 1: Comparison: GLPG1690 600 mg vs Placebo; Test type: Superiority; LS mean difference = 3.7, 95% CI 2-sided [-11.5 to 19.0] — The treatment effect was determined by using estimated least square mean difference between each active treatment group and placebo from the mixed model
Statistical Analysis 2: Comparison: GLPG1690 200 mg vs Placebo; Test type: Superiority; LS mean difference = 2.9, 95% CI 2-sided [-11.1 to 16.8] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Percentage of Participants With All Cause Hospitalization Until EoS
Description: Percentage of participants with all cause hospitalization was reported for this measure.
Time Frame: Up to EoS (week 121)
Population: Full Analysis Set - Efficacy
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 169 | 171 | 164
Percentage of participants | 18.3 | 21.6 | 18.9
Statistical Analysis 1: Comparison: GLPG1690 600 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.65 to 1.78] — Hazard ratio and 95% confidence interval originated from a Cox proportional hazards model for time to first all cause hospitalization
Statistical Analysis 2: Comparison: GLPG1690 200 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.76 to 1.98] — [estimate comment as in outcome 8, analysis 1]

9. Secondary Outcome: Percentage of Participants With Respiratory Related Mortality Until EoS
Description: Percentage of participants with respiratory related mortality until EoS were reported for this study.
Time Frame: Up to EoS (week 121)
Population: Full Analysis Set - Efficacy
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 169 | 171 | 164
Percentage of participants | 3.6 | 4.1 | 1.8

10. Secondary Outcome: Percentage of Participants Hospitalized for Non-elective Lung Transplant Until EoS
Description: Percentage of Participants who were hospitalized for Non-elective lung transplant were reported for this measure.
Time Frame: Up to EoS (week 121)
Population: Full Analysis Set - Efficacy
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 169 | 171 | 164
Percentage of participants | 0.0 | 0.0 | 0.0

11. Secondary Outcome: Percentage of Participants With Acute Idiopathic Pulmonary Fibrosis (IPF) Exacerbation Until EoS
Description: Percentage of participants with acute IPF exacerbation until EoS were reported for this measure.
Time Frame: Up to EoS (week 121)
Population: Full Analysis Set - Efficacy
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 169 | 171 | 164
Percentage of participants | 4.7 | 4.7 | 3.7
Statistical Analysis 1: Comparison: GLPG1690 600 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.44 to 3.81] — Hazard ratio and 95% confidence interval originated from a Cox proportional hazards model for time to first acute IPF exacerbation
Statistical Analysis 2: Comparison: GLPG1690 200 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.42 to 3.50] — [estimate comment as in outcome 11, analysis 1]

12. Secondary Outcome: Percentage of Participants With All Cause Mortality or Hospitalization for Non-elective Lung Transplant Until EoS
Description: Percentage of participants with all-cause mortality or hospitalization for non-elective lung transplant were reported for this measure.
Time Frame: Up to EoS (week 121)
Population: FAS - EF with available data at specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 161 | 171 | 164
Percentage of participants | 7.1 | 4.7 | 4.9
Statistical Analysis 1: Comparison: GLPG1690 600 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.64, 95% CI 2-sided [0.66 to 4.08] — Hazard ratio and 95% confidence interval originated from a Cox proportional hazards model for time to first all cause mortality or hospitalization for non-elective lung transplant
Statistical Analysis 2: Comparison: GLPG1690 200 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.36 to 2.61] — [estimate comment as in outcome 12, analysis 1]

13. Secondary Outcome: Percentage of Participants With All Cause Mortality, Hospitalization for Non-elective Lung Transplant or Hospitalization for Qualifying for Lung Transplant Until EoS
Description: Percentage of participants with all-cause mortality or hospitalization for non-elective lung transplant or hospitalization for qualifying for lung transplant were reported for this measure.
Time Frame: Up to EoS (week 121)
Population: Full Analysis Set - Efficacy
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 169 | 171 | 164
Percentage of participants | 7.1 | 4.7 | 4.9
Statistical Analysis 1: Comparison: GLPG1690 600 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.64, 95% CI 2-sided [0.66 to 4.08] — Hazard ratio and 95% confidence interval originated from a Cox proportional hazards model for time to first all cause mortality, hospitalization for non-elective lung transplant or hospitalization for qualifying for lung transplant
Statistical Analysis 2: Comparison: GLPG1690 200 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.36 to 2.61] — [estimate comment as in outcome 13, analysis 1]

14. Secondary Outcome: Percentage of Participants With All-Cause Mortality or Hospitalization That Meets >=10% Absolute Decline in %FVC or Respiratory-Related Hospitalization Until EoS
Description: Percentage of participants with all-cause mortality or respiratory related hospitalization that meets >=10% absolute decline in %FVC or respiratory-related hospitalization were reported for this measure.
Time Frame: Up to EoS (week 121)
Population: Full Analysis Set - Efficacy
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 169 | 171 | 164
Percentage of participants | 13.6 | 11.1 | 14.0
Statistical Analysis 1: Comparison: GLPG1690 600 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.59 to 1.91] — Hazard ratio and 95% confidence interval originated from a Cox proportional hazards model for time to first all-cause mortality or hospitalization that meets >=10% absolute decline in %FVC or respiratory-related hospitalization
Statistical Analysis 2: Comparison: GLPG1690 200 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.43 to 1.46] — [estimate comment as in outcome 14, analysis 1]

15. Secondary Outcome: Percentage of Participants With All-Cause Mortality or Respiratory-Related Hospitalizations Until EoS
Description: Percentage of participants with all-cause mortality or respiratory related hospitalization were reported for this measure.
Time Frame: Up to EoS (week 121)
Population: Full Analysis Set - Efficacy
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 169 | 171 | 164
Percentage of participants | 13.6 | 11.1 | 14.0
Statistical Analysis 1: Comparison: GLPG1690 600 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.59 to 1.91] — Hazard ratio and 95% confidence interval originated from a Cox proportional hazards model for time to all-cause mortality or respiratory-related hospitalizations
Statistical Analysis 2: Comparison: GLPG1690 200 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.43 to 1.46] — [estimate comment as in outcome 15, analysis 1]

16. Secondary Outcome: FVC at Week 52
Description: as for outcome 1
Time Frame: Week 52
Population: FAS-EF with available data at specified time point.
Measure: Mean (Standard Error); unit: mL
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 82 | 97 | 94
mL | 2886.20 (83.969) | 2662.90 (79.056) | 3021.99 (78.415)

17. Secondary Outcome: Change From Baseline in FVC at Week 52
Description: as for outcome 1
Time Frame: Baseline, week 52
Population: FAS-EF with available data at specified time point.
Measure: Mean (Standard Error); unit: mL
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 82 | 97 | 94
mL | -145.94 (31.799) | -182.29 (30.286) | -133.24 (31.819)

18. Secondary Outcome: Percent Change From Baseline in FVC at Week 52
Description: as for outcome 1
Time Frame: Baseline, week 52
Population: FAS-EF with available data at specified time point.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 82 | 97 | 94
Percent change | -4.57 (0.992) | -6.46 (1.115) | -4.48 (0.978)

19. Secondary Outcome: FVC at Week 112
Description: as for outcome 1
Time Frame: Week 112
Population: FAS-EF with available data at specified time point. No participant was available for analysis at Week 112 for arm "GLPG1690 200 mg" and "Placebo".
Measure: Mean (Standard Error); unit: mL
Arm/Group | GLPG1690 600 mg
Number analyzed (Participants) | 2
mL | 3262.00 (15.000)

20. Secondary Outcome: Change From Baseline in FVC at Week 112
Description: as for outcome 1
Time Frame: Baseline, week 112
Population: FAS - EF with available data at specified time point. No participant was available for analysis at Week 112 for arms "GLPG1690 200 mg" and "Placebo".
Measure: Mean (Standard Error); unit: mL
Arm/Group | GLPG1690 600 mg
Number analyzed (Participants) | 2
mL | -55.75 (277.750)

21. Secondary Outcome: Percent Change From Baseline in FVC at Week 112
Description: as for outcome 1
Time Frame: Baseline, week 112
Population: as for outcome 20
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | GLPG1690 600 mg
Number analyzed (Participants) | 2
Percent change | -0.95 (8.288)

22. Secondary Outcome: Percentage of Participants With Absolute Categorical Change From Baseline in Percent FVC at Week 52: FVC Change Within ≤5
Description: as for outcome 1
Time Frame: Baseline, week 52
Population: FAS - EF with available data at specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 82 | 97 | 94
Percentage of participants | 90.2 | 92.8 | 89.4

23. Secondary Outcome: Percentage of Participants With Absolute Categorical Change From Baseline in Percent FVC at Week 112: FVC Change Within ≤5
Description: as for outcome 1
Time Frame: Baseline, week 112
Population: as for outcome 20
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690 600 mg
Number analyzed (Participants) | 2
Percentage of participants | 50.0

24. Secondary Outcome: Percentage of Participants With Absolute Categorical Change From Baseline in Percent FVC at Week 52: FVC Change Within ≤10
Description: as for outcome 1
Time Frame: Baseline, week 52
Population: FAS - EF with available data at specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 82 | 97 | 94
Percentage of participants | 97.6 | 97.9 | 96.8

25. Secondary Outcome: Percentage of Participants With Absolute Categorical Change From Baseline in Percent FVC at Week 112: FVC Change Within ≤10
Description: as for outcome 1
Time Frame: Baseline, week 112
Population: as for outcome 20
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690 600 mg
Number analyzed (Participants) | 2
Percentage of participants | 100

26. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: Safety was assessed by AEs, which included abnormalities identified during a medical test (example, laboratory tests, vital signs, electrocardiogram, etc.) if the abnormality induced clinical signs or symptoms, needed active intervention, interruption or discontinuation of study drug or was clinically significant. A Treatment emergent AE (TEAE) was defined as any AE that started or worsened after the first dose of study drug up to 30 days after the last dose of study drug. AEs were considered serious (SAEs) if the AE resulted in death, was life-threatening, resulted in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, resulted in congenital anomaly, or birth defect or required inpatient hospitalization or led to prolongation of hospitalization.
Time Frame: Baseline up to 30 days after the last dose (up to week 121)
Population: FAS consisted of all randomized participants who received at least 1 dose of investigational product.
Measure: Number; unit: Percentage of participants
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 174 | 175 | 174
Percentage of participants
  TEAEs | 78.7 | 84.6 | 84.5
  Serious TEAEs | 21.8 | 21.7 | 20.7

27. Secondary Outcome: Changes From Baseline Leicester Cough Questionnaire (LCQ) Total Score and Individual Domain Score at Week 52 and Week 100
Description: Cough was evaluated using the LCQ. The LCQ was a 19-item questionnaire split into three domains: physical, psychological, and social. Scores were calculated by domain (range from 1 to 7, higher scores indicated a better health status) and then the total score was calculated by adding the individual domain score. Total score ranged from 3 to 21, with higher scores indicated a better health status.
Time Frame: Baseline, week 52, week 100
Population: FAS - EF with available data at specified time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 89 | 104 | 97
Score on a scale
  Physical Score: Change at Week 52 | 0.024 (1.218) | -0.215 (0.966) | -0.151 (0.835)
  Physical Score: Change at Week 100: number analyzed (Participants) | 6 | 9 | 7
  Physical Score: Change at Week 100 | -0.208 (0.452) | -0.222 (1.200) | -0.286 (0.847)
  Psychological Score: Change at Week 52 | -0.122 (1.397) | -0.225 (1.204) | -0.044 (1.020)
  Psychological Score: Change at Week 100: number analyzed (Participants) | 6 | 9 | 7
  Psychological Score: Change at Week 100 | -0.595 (0.941) | -0.254 (0.892) | 0.367 (0.899)
  Social Score: Change at Week 52 | -0.065 (1.344) | -0.351 (1.147) | -0.052 (1.080)
  Social Score: Change at Week 100: number analyzed (Participants) | 6 | 9 | 7
  Social Score: Change at Week 100 | -0.458 (1.269) | -0.333 (1.237) | 0.321 (0.997)
  Total Score: Change at Week 52 | -0.163 (3.778) | -0.791 (3.028) | -0.247 (2.680)
  Total Score: Change at Week 100: number analyzed (Participants) | 6 | 9 | 7
  Total Score: Change at Week 100 | -1.262 (2.295) | -0.810 (0.9249) | 0.403 (2.497)

28. Secondary Outcome: Change From Baseline in Visual Analogue Score (VAS): Cough at Week 52 and Week 100
Description: Cough was assessed using VAS score, ranged from 0 (no cough) to 100 millimeter (mm) (worst possible cough).
Time Frame: Baseline, week 52, week 100
Population: FAS-EF with available data at specified time point
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 89 | 104 | 96
mm
  Change at Week 52 | 2.9 (27.9) | 3.2 (25.1) | 2.3 (27.3)
  Change at Week 100: number analyzed (Participants) | 6 | 9 | 7
  Change at Week 100 | 8.0 (23.1) | 0.3 (24.0) | 25.4 (39.1)

29. Secondary Outcome: Change From Baseline in Visual Analogue Score (VAS): Urge to Cough at Week 52 and Week 100
Description: Urge to Cough was assessed using VAS score, ranged from 0 (no urge to cough) to 100 mm (highest urge to cough).
Time Frame: Baseline, week 52, week 100
Population: FAS-EF with available data at specified time point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 89 | 104 | 96
mm
  Change at Week 52 | 1.8 (26.8) | 1.5 (23.2) | 1.1 (24.9)
  Change at Week 100: number analyzed (Participants) | 6 | 9 | 7
  Change at Week 100 | 5.7 (22.0) | -1.9 (24.8) | 24.3 (40.6)

30. Secondary Outcome: Change From Baseline in European Quality Of Life (EQ) VAS at Week 52 and Week 100
Description: EuroQol outcome measurements is a printed 20 cm VAS that appears somewhat like a thermometer, on which a score from 0 (worst imaginable health state or death) to 100 (best imaginable health state) was marked by the participant (or, when necessary, their proxy) with the scale in view.
Time Frame: Baseline, week 52, week 100
Population: FAS-EF with available data at specified time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 90 | 104 | 97
Score on a scale
  Change at Week 52 | -1.4 (16.2) | -6.1 (17.3) | -3.7 (16.5)
  Change at Week 100 | 7.2 (12.3) | -9.3 (25.2) | -2.1 (23.8)

31. Secondary Outcome: Change From Baseline in King's Brief Interstitial Lung Disease (K-BILD) at Week 52 and Week 100
Description: The K-BILD questionnaire was specifically developed to analyze the health status of participants with ILD. The questionnaire consists of 15 items (assessed by the participants on a scale ranging from 1 to 7, where 1 and 7 represent worst and best health status). Items are compiled into 3 domains: breathlessness and activities (range: 0-21), psychological (range: 0-34) , and chest symptoms (range: 0-8). To score the K-BILD, the Likert response scale weightings for individual items are combined and scores are transformed to a range of 0-100 by using logit values (higher scores indicate better health status).
Time Frame: Baseline, week 52, week 100
Population: FAS-EF with available data at specified time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 89 | 104 | 96
Score on a scale
  Breathlessness and Activities Score: Change at Week 52 | -0.256 (20.896) | -5.031 (13.512) | -4.545 (15.250)
  Breathlessness and Activities Score: Change at Week 100: number analyzed (Participants) | 6 | 9 | 7
  Breathlessness and Activities Score: Change at Week 100 | 1.417 (19.427) | -9.733 (15.973) | -3.843 (19.788)
  Psychological Score: Change at Week 52 | 0.429 (18.240) | -2.583 (15.555) | -2.421 (17.049)
  Psychological Score: Change at Week 100 | -4.417 (30.117) | -6.478 (9.193) | -2.743 (10.930)
  Chest Symptoms Score: Change at Week 52 | -1.624 (20.367) | -2.095 (20.002) | -2.790 (20.052)
  Chest Symptoms Score: Change at Week 100: number analyzed (Participants) | 6 | 9 | 7
  Chest Symptoms Score: Change at Week 100 | 0.850 (13.686) | -2.667 (19.951) | -3.371 (16.023)
  Total Score: Change at Week 52 | -0.276 (13.690) | -2.306 (10.398) | -2.484 (10.863)
  Total Score: Change at Week 100: number analyzed (Participants) | 6 | 9 | 7
  Total Score: Change at Week 100 | -0.383 (15.090) | -5.444 (7.726) | -2.371 (10.520)

32. Secondary Outcome: Area Under The Concentration Time Curve (AUC) of Ziritaxtestat
Description: Area under the concentration time curve of ziritaxtestat was reported.
Time Frame: Sparse samples collected on day 1 pre-dose, day 85 post-dose, day 237 post-dose, day 183 pre-dose, day 365 pre-dose
Population: Pharmacokinetic Analysis Set: All randomized participants who received at least one dose of IP and for whom evaluable PK data were available.
Measure: Median (90% Confidence Interval); unit: Nanogram * milliliter per hour (ng*mL/h)
Groups:
- GLPG1690 200 mg: Participants received GLPG1690 (ziritaxestat) 200 mg as film-coated tablet for oral use once daily (mean GLPG1690 exposure was up to 356.0 days).
- GLPG1690 600 mg: Participants received GLPG1690 (ziritaxestat) 600 mg, film-coated tablets orally once daily (mean GLPG1690 exposure was up to 325.3 days).
- GLPG1690 200 mg/Nintedanib: Participants received GLPG1690 (ziritaxestat) 200 mg, film-coated tablets orally once daily (mean GLPG1690 exposure was up to 325.3 days) in addition to local standard of care. Standard of care included nintedanib at a stable dose for at least 2 months before screening, and during screening;
- GLPG1690 600 mg/Nintedanib: Participants received GLPG1690 (ziritaxestat) 600 mg, film-coated tablets orally once daily (mean GLPG1690 exposure was up to 325.3 days) in addition to local standard of care. Standard of care included nintedanib at a stable dose for at least 2 months before screening, and during screening;
- GLPG1690 200 mg/Pirfenidone: Participants received GLPG1690 (ziritaxestat) 200 mg, film-coated tablets orally once daily (mean GLPG1690 exposure was up to 325.3 days) in addition to local standard of care. Standard of care included pirfenidone at a stable dose for at least 2 months before screening, and during screening;
- GLPG1690 600 mg/Pirfenidone: Participants received GLPG1690 (ziritaxestat) 600 mg, film-coated tablets orally once daily (mean GLPG1690 exposure was up to 325.3 days) in addition to local standard of care. Standard of care included pirfenidone at a stable dose for at least 2 months before screening, and during screening;
Arm/Group | GLPG1690 200 mg | GLPG1690 600 mg | GLPG1690 200 mg/Nintedanib | GLPG1690 600 mg/Nintedanib | GLPG1690 200 mg/Pirfenidone | GLPG1690 600 mg/Pirfenidone
Number analyzed (Participants) | 24 | 18 | 24 | 26 | 30 | 27
Nanogram * milliliter per hour (ng*mL/h) | 10367 [7960.4 to 12773.6] | 51136 [40132.9 to 62139.1] | 7095 [6411.3 to 7778.7] | 33796 [29021.56 to 38570.44] | 6375 [5907.28 to 6842.72] | 21188 [16847.76 to 25528.24]

33. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ziritaxtestat
Description: Maximum Observed Plasma Concentration of Ziritaxtestat was reported.
Time Frame: Sparse samples collected on day 1 pre-dose, day 85 post-dose, day 237 post-dose, day 183 pre-dose, day 365 pre-dose
Population: Pharmacokinetic Analysis Set
Measure: Median (90% Confidence Interval); unit: Nanogram per milliliter (ng/mL)
Arm/Group | GLPG1690 200 mg | GLPG1690 600 mg | GLPG1690 200 mg/Nintedanib | GLPG1690 600 mg/Nintedanib | GLPG1690 200 mg/Pirfenidone | GLPG1690 600 mg/Pirfenidone
Number analyzed (Participants) | 24 | 18 | 24 | 26 | 30 | 27
Nanogram per milliliter (ng/mL) | 864 [721.42 to 1006.58] | 3962 [3330.09 to 4593.91] | 583 [541.55 to 624.45] | 2686 [2414.7 to 2957.3] | 591 [556.46 to 625.54] | 2009 [1692.94 to 2325.06]

34. Secondary Outcome: Change From Baseline in Total Distance Walked in Six-minute Walk Test (6MWT) at Week 52 and Week 100
Description: The 6-MWT depicted the total distance covered by a participant during 6 minutes of walking.
Time Frame: Baseline, week 52, week 100
Population: FAS - EF with available data at specified time point.
Measure: Mean (Standard Error); unit: Meter
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 67 | 73 | 80
Meter
  Change at Week 52 | -36.34 (7.805) | -15.65 (9.865) | -34.75 (11.546)
  Change at Week 100: number analyzed (Participants) | 3 | 2 | 2
  Change at Week 100 | -83.00 (17.521) | -79.00 (13.00) | -137.87 (93.135)

35. Secondary Outcome: Change From Baseline in Diffusing Capacity of Lung for Carbon Monoxide (DLCO) (Corrected for Hemoglobin [Hb]) at Week 52 and Week 100
Description: Change from baseline in DLCO (percent predicted hemoglobin level corrected) was reported for this measure.mmol/min/kPa: Millimole per minute per kilopascal
Time Frame: Baseline, week 52, week 100
Population: FAS - EF with available data at specified time point.
Measure: Mean (Standard Error); unit: mmol/min/kPa
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
Number analyzed (Participants) | 60 | 77 | 73
mmol/min/kPa
  Change at Week 52 | -0.640 (0.1205) | -0.137 (0.1288) | -0.193 (0.0907)
  Change at Week 100: number analyzed (Participants) | 3 | 1 | 2
  Change at Week 100 | -0.215 (0.6737) | -1.670 | -2.134 (1.9836)

ADVERSE EVENTS:
Time Frame: Baseline Up to 30 days after the last dose (Up to week 121)
Description: FAS consisted of all randomized participants who received at least 1 dose of investigational product.
Arm/Group | GLPG1690 600 mg | GLPG1690 200 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 12/174 | 8/175 | 8/174
Serious Adverse Events (participants affected / at risk) | 38/174 | 38/175 | 36/174
Other Adverse Events (participants affected / at risk) | 91/174 | 99/175 | 82/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLPG1690 600 mg (N=174) | GLPG1690 200 mg (N=175) | Placebo (N=174)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 2 (3)
Myocardial rupture (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial haemorrhage (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Femoral hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Drug intolerance (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1) | 2 (3)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 3 (6) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (3)
Pneumonia (Infections and infestations) | 4 (7) | 2 (3) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (3) | 0 (0) | 1 (1)
Platelet morphology abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Cubital tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Limbic encephalitis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Device loosening (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (3) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (5) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 12 (20) | 7 (16) | 12 (19)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 2 (2)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLPG1690 600 mg (N=174) | GLPG1690 200 mg (N=175) | Placebo (N=174)
Diarrhoea (Gastrointestinal disorders) | 51 (111) | 40 (84) | 20 (33)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 (10) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 16 (18) | 14 (20) | 10 (14)
Fatigue (General disorders) | 10 (10) | 9 (12) | 6 (7)
Bronchitis (Infections and infestations) | 8 (10) | 11 (13) | 4 (4)
Nasopharyngitis (Infections and infestations) | 11 (14) | 7 (10) | 10 (11)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 12 (15) | 11 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 9 (13) | 9 (10)
Dizziness (Nervous system disorders) | 8 (10) | 4 (4) | 9 (9)
Headache (Nervous system disorders) | 9 (14) | 13 (15) | 10 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 21 (25) | 16 (18)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 17 (25) | 10 (10)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 12 (15) | 13 (18)

LIMITATIONS AND CAVEATS:
This Study was prematurely terminated based on recommendations of the Independent Data Monitoring Committee.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review and approve any results of the study or abstracts for professional meetings prepared by the investigator(s). Published data must not compromise the objectives of the study. Data from individual study centers in multicenter studies must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/62/NCT03711162/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT03711162/SAP_001.pdf